CLINICAL TRIAL: NCT00517530
Title: An Open-label, Multicentre, Nonrandomized, Dose-escalating Phase I/II Study, With a Randomized Phase II Part, to Investigate the Safety and Tolerability of RO5072759 Given as Monotherapy in Patients With CD20+ Malignant Disease.
Brief Title: A Dose-Escalating Study of Obinutuzumab in Patients With B-lymphocyte Antigen (CD20+) Malignant Disease (GAUGUIN)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO20999; 2007-001103-37 (EudraCT Number)
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Phase I, NHL (Experimental): Participants in this NHL arm received multiple ascending doses between 50 and 2000 mg via intravenous infusion of obinutuzumab.
  Interventions: Drug: Obinutuzumab
- Phase I, CLL (Experimental): Participants in this CLL arm received multiple ascending doses between 400 and 2000 mg via intravenous infusion of obinutuzumab.
  Interventions: Drug: Obinutuzumab
- 400/400 mg - Phase II, iNHL (Experimental): Participants in this iNHL arm received an intravenous infusion of obinutuzumab 400 mg on Days 1 and 8 of Cycle 1 and obinutuzumab 400 mg on Day 1 of Cycles 2-8 for a maximum of 8 cycles and 9 infusions. Each cycle was 21 days.
  Interventions: Drug: Obinutuzumab
- 1600/800 mg - Phase II, iNHL (Experimental): Participants in this iNHL arm received an intravenous infusion of obinutuzumab 1600 mg on Days 1 and 8 of Cycle 1 and obinutuzumab 800 mg on Day 1 of Cycles 2-8 for a maximum of 8 cycles and 9 infusions. Each cycle was 21 days.
  Interventions: Drug: Obinutuzumab
- 400/400 mg - Phase II, aNHL (Experimental): Participants in this aNHL arm received an intravenous infusion of obinutuzumab 400 mg on Days 1 and 8 of Cycle 1 and obinutuzumab 400 mg on Day 1 of Cycles 2-8 for a maximum of 8 cycles and 9 infusions. Each cycle was 21 days.
  Interventions: Drug: Obinutuzumab
- 1600/800 mg - Phase II, aNHL (Experimental): Participants in this aNHL arm received an intravenous infusion of obinutuzumab 1600 mg on Days 1 and 8 of Cycle 1 and obinutuzumab 800 mg on Day 1 of Cycles 2-8 for a maximum of 8 cycles and 9 infusions. Each cycle was 21 days.
  Interventions: Drug: Obinutuzumab
- 1000/1000 mg - Phase II, CLL (Experimental): Participants in this CLL arm received an intravenous infusion of obinutuzumab 1000 mg on Days 1, 8, and 15 of Cycle 1 and obinutuzumab 1000 mg on Day 1 of Cycles 2-8 for a maximum of 8 cycles and 10 infusions. Each cycle was 21 days.
  Interventions: Drug: Obinutuzumab
- Retreated Participants (Experimental): Participants who might benefit from retreatment who were allowed to be treated again via intravenous infusion of obinutuzumab at the request of the investigator.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab was provided in single-dose glass vials as a freeze-dried powder.
  Other Names: RO5072759; GA101

SUMMARY:
The primary objective for the phase I part of the study is to investigate the safety and tolerability of escalating intravenous (IV) doses of obinutuzumab given as monotherapy in participants with CD20+ (tumor-infiltrating lymphocytic) Malignant Disease, including B-cell chronic lymphocytic leukemia (CLL) and Non-Hodgkin's Lymphoma (NHL). The primary objective for the phase II part of the study is to investigate the efficacy and safety of one dose of obinutuzumab in participants with relapsed/refractory CLL and NHL that is, in turn, either indolent (iNHL) or aggressive (aNHL).

It is an open label dose escalating study in phase I and open label in phase II, but the two doses in iNHL & aNHL are randomized (to high or low dose of the same open label treatment). CLL was not randomized as only one dose level was used.

Participants with a response who might gain additional benefit from being treated again in the opinion of the investigator may be enrolled in a Retreatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age;
* Phase 1 only: CD20+ malignant disease (B-cell lymphoma or B-CLL);
* Phase 2 only: relapsed or refractory indolent NHL, relapsed or refractory aggressive NHL or relapsed or refractory B-CLL
* Have a clinical indication for treatment as determined by the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy >12 weeks

Exclusion Criteria:

* Prior use of any investigational antibody therapy or other agent within 6 months of study start;
* Prior use of any anti-cancer vaccine;
* Prior use of standard anti-lymphoma/leukemia therapy or radiation therapy within 4 weeks of enrollment;
* Prior use of MabThera (rituximab) within 8 weeks of study entry;
* Prior administration of radioimmunotherapy 3 months prior to study entry;
* Central nervous system (CNS) lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- France (14):
  - Créteil
  - Le Mans
  - Lille
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rennes
  - Rouen
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
- Cologne, Germany

REFERENCES:
- [Derived] Gibiansky E, Gibiansky L, Buchheit V, Frey N, Brewster M, Fingerle-Rowson G, Jamois C. Pharmacokinetics, exposure, efficacy and safety of obinutuzumab in rituximab-refractory follicular lymphoma patients in the GADOLIN phase III study. Br J Clin Pharmacol. 2019 Sep;85(9):1935-1945. doi: 10.1111/bcp.13974. Epub 2019 Jul 12. PMID 31050355
- [Derived] Cartron G, Hourcade-Potelleret F, Morschhauser F, Salles G, Wenger M, Truppel-Hartmann A, Carlile DJ. Rationale for optimal obinutuzumab/GA101 dosing regimen in B-cell non-Hodgkin lymphoma. Haematologica. 2016 Feb;101(2):226-34. doi: 10.3324/haematol.2015.133421. Epub 2015 Dec 11. PMID 26659915
- [Derived] Cartron G, de Guibert S, Dilhuydy MS, Morschhauser F, Leblond V, Dupuis J, Mahe B, Bouabdallah R, Lei G, Wenger M, Wassner-Fritsch E, Hallek M. Obinutuzumab (GA101) in relapsed/refractory chronic lymphocytic leukemia: final data from the phase 1/2 GAUGUIN study. Blood. 2014 Oct 2;124(14):2196-202. doi: 10.1182/blood-2014-07-586610. Epub 2014 Aug 20. PMID 25143487
- [Derived] Morschhauser FA, Cartron G, Thieblemont C, Solal-Celigny P, Haioun C, Bouabdallah R, Feugier P, Bouabdallah K, Asikanius E, Lei G, Wenger M, Wassner-Fritsch E, Salles GA. Obinutuzumab (GA101) monotherapy in relapsed/refractory diffuse large b-cell lymphoma or mantle-cell lymphoma: results from the phase II GAUGUIN study. J Clin Oncol. 2013 Aug 10;31(23):2912-9. doi: 10.1200/JCO.2012.46.9585. Epub 2013 Jul 8. PMID 23835718
- [Derived] Salles GA, Morschhauser F, Solal-Celigny P, Thieblemont C, Lamy T, Tilly H, Gyan E, Lei G, Wenger M, Wassner-Fritsch E, Cartron G. Obinutuzumab (GA101) in patients with relapsed/refractory indolent non-Hodgkin lymphoma: results from the phase II GAUGUIN study. J Clin Oncol. 2013 Aug 10;31(23):2920-6. doi: 10.1200/JCO.2012.46.9718. Epub 2013 Jul 8. PMID 23835715
- [Derived] Salles G, Morschhauser F, Lamy T, Milpied N, Thieblemont C, Tilly H, Bieska G, Asikanius E, Carlile D, Birkett J, Pisa P, Cartron G. Phase 1 study results of the type II glycoengineered humanized anti-CD20 monoclonal antibody obinutuzumab (GA101) in B-cell lymphoma patients. Blood. 2012 May 31;119(22):5126-32. doi: 10.1182/blood-2012-01-404368. Epub 2012 Mar 19. PMID 22431570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Different patients were recruited into Phase I and Phase II, and analyzed separately based on their disease. In this adaptive trial design, some of those same patients were included in follow-up even if they did not complete treatment, and 13 who had initially responded to treatment but subsequently progressed were retreated.
Groups:
- 50-2000 mg Phase I, NHL; 400-2000 mg Phase I, CLL; 400/400 mg - Phase II, iNHL; 1600/800 mg - Phase II, iNHL; 400/400 mg - Phase II, aNHL; 1600/800 mg - Phase II, aNHL; 1000/1000 mg - Phase II, CLL: Obinutuzumab intravenous infusion
Period: Overall Study
Arm/Group | 50-2000 mg Phase I, NHL | 400-2000 mg Phase I, CLL | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Started | 21 | 13 | 18 | 22 | 21 | 19 | 20
Completed Treatment | 11 | 13 | 13 | 18 | 9 | 9 | 13
Started Follow-up | 20 | 13 | 17 | 21 | 17 | 16 | 19
Completed Follow-up | 2 | 0 | 0 | 1 | 0 | 0 | 1
Retreated Population | 2 | 2 | 1 | 4 | 2 | 2 | 0
Completed | 2 | 0 | 0 | 1 | 1 | 0 | 1
Not Completed | 19 | 13 | 18 | 21 | 20 | 19 | 19

BASELINE CHARACTERISTICS:
Population: Safety population: All enrolled participants who had received at least 1 dose of obinutuzumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | 50-2000 mg Phase I, NHL | 400-2000 mg Phase I, CLL | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL | Total
Number analyzed (Participants) | 21 | 13 | 18 | 22 | 21 | 19 | 20 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 14 | 14 | 6 | 7 | 11 | 70
  >=65 years | 10 | 6 | 4 | 8 | 15 | 12 | 9 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 6 | 9 | 8 | 5 | 8 | 52
  Male | 9 | 9 | 12 | 13 | 13 | 14 | 12 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Dose-limiting Toxicity in Phase I of the Study
Description: Dose-limiting toxicities were defined as obinutuzumab-related adverse events occurring within the first 28 days of each administration of obinutuzumab, with the exception of B-cell depletion and lymphopenia which are expected outcomes of treatment with obinutuzumab.
Time Frame: Baseline to 28 days after the last infusion of obinutuzumab (up to 6 months)
Population: Safety population: All enrolled participants in Phase I, who had received at least 1 dose of obinutuzumab by 6 months.
Measure: Number; unit: percentage of participants
Groups:
- 50/100 mg - Phase I, NHL; 100/200 mg - Phase I, NHL; 200/400 mg - Phase I, NHL; 400/800 mg - Phase I, NHL; 800/1200 mg - Phase I, NHL; 1200/2000 mg - Phase I, NHL; 1600/800 mg - Phase I, NHL; 400/800 mg - Phase I, CLL; 800/1200 mg - Phase I, CLL; 1200/2000 mg - Phase I, CLL; 1000/1000 mg - Phase I, CLL: Obinutuzumab intravenous infusion
Arm/Group | 50/100 mg - Phase I, NHL | 100/200 mg - Phase I, NHL | 200/400 mg - Phase I, NHL | 400/800 mg - Phase I, NHL | 800/1200 mg - Phase I, NHL | 1200/2000 mg - Phase I, NHL | 1600/800 mg - Phase I, NHL | 400/800 mg - Phase I, CLL | 800/1200 mg - Phase I, CLL | 1200/2000 mg - Phase I, CLL | 1000/1000 mg - Phase I, CLL
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Best Overall Response in Phase II of the Study
Description: Best overall response (BOR) was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Time Frame: by Cutoff Date: 31 March 2012 (within 3 years, 4 months)
Population: Safety population: All enrolled participants in Phase II, who had received at least 1 dose of obinutuzumab.
Measure: Number; unit: percentage of participants
Arm/Group | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Number analyzed (Participants) | 18 | 22 | 21 | 19 | 20
percentage of participants | 33.3 | 63.6 | 23.8 | 36.8 | 30.0

3. Secondary Outcome: Percentage of Participants With Complete Response (CR/CRu/CRi) in Phase II of the Study
Description: A complete response was defined as the disappearance of all evidence of disease (NHL) and symptoms; normalization of biochemical abnormalities (NHL); regression of lymph nodes and nodal masses to normal size; decrease of nodes in the sum of the products of the greatest diameters (SPD); regression in size of the spleen and/or liver, should not be palpable, and disappearance of nodules related to lymphoma (CLL). Complete/unconfirmed (CRu) response includes NHL patients with one or more of the following: 1) a residual lymph node mass greater than 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the SPD; 2) Indeterminate bone marrow (increased number or size of aggregates without cytologic or architectural atypia). Complete Response with Incomplete Bone Marrow Recovery (CRi) was measured only in patients with CLL.
Time Frame: by Cutoff Date: 31 March 2012 (within 3 years, 4 months)
Measure: Number; unit: percentage of participants
Arm/Group | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Number analyzed (Participants) | 18 | 22 | 21 | 19 | 20
percentage of participants
  CR | 5.6 | 13.6 | 9.5 | 15.8 | 5.0
  CRu | 5.6 | 9.1 | 4.8 | 0.0 | NA — CRu was measured only in participants with NHL
  CRi | NA — CRi was measured only in participants with CLL | NA — CRi was measured only in participants with CLL | NA — CRi was measured only in participants with CLL | NA — CRi was measured only in participants with CLL | 0.0

4. Secondary Outcome: Percentage of Participants With Partial Response (PR) in Phase II of the Study
Description: A PR was defined as a >=50% decrease in SPD of the 6 largest nodes or nodal masses; no increase in size of other nodes, liver, or spleen; regression of splenic and hepatic nodules by >=50% in their SPD or, for single nodules, in the long axis (CLL only); and no new disease sites.
Time Frame: by Cutoff Date: 31 March 2012 (within 3 years, 4 months)
Measure: Number; unit: percentage of participants
Arm/Group | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Number analyzed (Participants) | 18 | 22 | 21 | 19 | 20
percentage of participants | 22.2 | 40.9 | 9.5 | 21.1 | 25.0

5. Secondary Outcome: Progression-free Survival (PFS) in Phase II of the Study
Description: PFS was defined as the time from start of treatment to disease progression (PD) or death due to any cause, whichever occurred first. For non-Hodgkin's lymphoma participants, PD was defined as >= 50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal node for participants with a partial response or non-responders or the appearance of any new lesion during or at the end of therapy. For chronic lymphocytic leukemia participants, PD was defined as: (1) A >= 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or the size of other lesions (eg, splenic or hepatic nodules); a lymph node with a short axis of < 1.0 cm must increase by >= 50% and to a size of 1.5×1.5 cm or > 1.5 cm in the longest axis. (2) Appearance of any new lesion > 1 cm in the short axis. (4) A new site that is positron emission tomography (PET)-positive with histological confirmation.
Time Frame: by the end of the follow-up period in Phase II of the study (within 3 years, 4 months)
Population: Safety population: All enrolled participants in Phase II, who had received at least 1 dose of obinutuzumab.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Number analyzed (Participants) | 18 | 22 | 21 | 19 | 20
days | 182 [106 to 526] | 361 [343 to 678] | 78 [42 to 260] | 83 [43 to 339] | 324 [217 to 357]

6. Secondary Outcome: Duration of Response by Disease Type in Phase II of the Study
Description: Duration of complete response was defined as the time from the first complete or partial response until disease progression (PD) or death, whichever occurred first. For non-Hodgkin's lymphoma participants, PD was defined as >= 50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal node for participants with a partial response or non-responders or the appearance of any new lesion during or at the end of therapy. For chronic lymphocytic leukemia participants, PD was defined as: (1) A >= 50% increase from nadir in the SPD of any previously involved nodes, or in a single involved node, or the size of other lesions (eg, splenic or hepatic nodules); a lymph node with a short axis of < 1.0 cm must increase by >= 50% and to a size of 1.5×1.5 cm or > 1.5 cm in the longest axis. (2) Appearance of any new lesion > 1 cm in the short axis. (4) A new site that is PET-positive with histological confirmation.
Time Frame: by the end of the follow-up period in Phase II of the study (within 3 years, 4 months)
Population: Safety population: All enrolled participants in Phase II, who had received at least 1 dose of obinutuzumab. Data reported for each disease cohort.
Measure: Median (Full Range); unit: days
Groups:
- Phase II, iNHL; Phase II, aNHL: Obinutuzumab intravenous infusion at 400/400 mg and 1600/800 mg
- Phase II, CLL: Obinutuzumab intravenous infusion at 1000/1000 mg
Arm/Group | Phase II, iNHL | Phase II, aNHL | Phase II, CLL
Number analyzed (Participants) | 20 | 12 | 6
days | 523 [23 to 952] | 298 [95 to 929] | 272.5 [23 to 794]

7. Secondary Outcome: Participants With Event-Free Survival (EFS) in Phase II of the Study
Description: EFS is defined as the time from start of treatment to disease progression/relapse, death or, in case of early withdrawal from the treatment period, the (end) date of last dose, whatever comes first.
Time Frame: by the end of the follow-up period in Phase II of the study (within 3 years, 4 months)
Measure: Number; unit: participants
Arm/Group | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Number analyzed (Participants) | 18 | 22 | 21 | 19 | 20
participants | 5 | 6 | 2 | 3 | 4

8. Secondary Outcome: Pharmacodynamics: Participants With Peripheral B-cell Recovery After Having Had Depletion at End of Treatment During Phase II of the Study
Description: B-cell depletion was defined in two ways: definition 1 - decrease below 5% baseline level and definition 2 - decrease below 0.04 x 109/L. B-cell recovery was defined in two ways: definition 1 - return to at least 50% of baseline level and definition 2 - return to at least 0.08 x 109/L.
Time Frame: by the end of Phase II (within 3 years, 4 months)
Population: Participants analyzed include those with B-cell depletion at the end of treatment (N), with assessments (n) at each time point.
Measure: Number; unit: participants
Arm/Group | 400/400 mg - Phase II, iNHL | 1600/800 mg - Phase II, iNHL | 400/400 mg - Phase II, aNHL | 1600/800 mg - Phase II, aNHL | 1000/1000 mg - Phase II, CLL
Number analyzed (Participants) | 16 | 21 | 21 | 19 | 16
participants
  within 6 months (n=11,19,11,12,13) | 0 | 0 | 0 | 0 | 3
  within 9 months (n=8,17,6,5,10) | 0 | 0 | 0 | 1 | 0
  within 12 months (n=5,16,4,5,9) | 0 | 2 | 1 | 0 | 3
  within 18 months (n=4,13,3,3,8) | 0 | 1 | 0 | 1 | 2
  within 24 months (n=3,10,2,3,5) | 2 | 2 | 1 | 0 | 2
  after 24 months (n=3,4,1,2,0) | 1 | 0 | 0 | 1 | 0

9. Secondary Outcome: Percentage of Retreated Participants With Response
Description: Patients who might benefit from retreatment were allowed to be treated again at the request of the investigator.
Time Frame: by Cutoff Date: 25 November 2013 (within 4 years, 2 months)
Population: Retreated participants
Measure: Number; unit: percentage of participants
Groups:
- Retreated Participants: Obinutuzumab intravenous infusion
Arm/Group | Retreated Participants
Number analyzed (Participants) | 13
percentage of participants
  Best overall response | 62
  Complete response | 23
  Partial response | 38

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Obinutuzumab in NHL Participants
Description: Obinutuzumab serum pharmacokinetic (PK) parameters in NHL participants following ascending doses.
Time Frame: at Cycle 1 Day 1, Cycle 1 Day 8 and Cycle 8 (over 168 days)
Population: Pharmacokinetics (PK)- evaluable population at the given dose (e.g., 3 or more participants at any of the given time points). Other doses did not have a PK-evaluable population, so were not included in the table of results. Due to the limited sampling schedule derived PK parameters could not be accurately obtained during Cycle 1 and Cycle 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µm/ml*day
Groups:
- 400 mg - Phase I, NHL; 800 mg - Phase I, NHL; 1200 mg - Phase I, NHL; 2000 mg - Phase I, NHL: Obinutuzumab intravenous infusion
Arm/Group | 400 mg - Phase I, NHL | 800 mg - Phase I, NHL | 1200 mg - Phase I, NHL | 2000 mg - Phase I, NHL
Number analyzed (Participants) | 4 | 6 | 6 | 6
µm/ml*day
  Cycle 1 Day 1 (n=4,6,6,0) | 134 (27.1) | 234 (63.1) | 307 (30.6) | NA (NA) — n=0
  Cycle 1 Day 8 (n=0,4,6,6) | NA (NA) — n=0 | 367 (24.2) | 449 (26.4) | 714 (28.6)
  Cycle 8 (n=0,5,5,5) | NA (NA) — n=0 | 698 (65.4) | 1070 (62.6) | 1380 (66.1)

11. Secondary Outcome: Area Under the Concentration-time Curve of Obinutuzumab Administered on Day 1 of Cycle 1 in Phase I of the Study
Description: Blood samples were taken on Day 1 (pre-infusion, end of infusion, 3-6 hours post-infusion) of Cycle 1. Nonlinear mixed-effects modeling (with NONMEM software) was used to analyze the pooled samples for dose-concentration-time data of obinutuzumab.
Time Frame: Day 1 of Cycle 1
Population: Pharmacokinetics (PK)- evaluable population at the given dose (e.g., 3 or more participants). Other doses did not have a PK-evaluable population, so were not included in the table of results. Due to the limited sampling schedule derived PK parameters could not be accurately obtained during Cycle 1 and Cycle 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µm/ml*day
Arm/Group | 400 mg - Phase I, NHL | 800 mg - Phase I, NHL | 1200 mg - Phase I, NHL | 2000 mg - Phase I, NHL
Number analyzed (Participants) | 4 | 6 | 6 | 3
µm/ml*day | 459 (64.7) | 993 (30.5) | 1057 (60.5) | 146 (49.6)

12. Other Pre Specified Outcome: Maximum Plasma Concentration (Cmax) of Obinutuzumab in CLL Patients
Time Frame: at Cycle 1 Day 1, Cycle 1 Day 8 and Cycle 8 (over 168 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/mL
Groups:
- 400 mg - Phase I, CLL; 800 mg - Phase I, CLL; 1200 mg - Phase I, CLL; 2000 mg - Phase I, CLL: Obinutuzumab intravenous infusion
Arm/Group | 400 mg - Phase I, CLL | 800 mg - Phase I, CLL | 1200 mg - Phase I, CLL | 2000 mg - Phase I, CLL
Number analyzed (Participants) | 3 | 4 | 4 | 4
micrograms/mL
  Cycle 1 Day 1 (n=3,3,3,0) | 216 (34.1) | 210 (74.0) | 307 (21.4) | NA (NA) — n=0
  Cycle 1 Day 8 (n=0,0,3,3) | NA (NA) — n=0 | NA (NA) — n=0 | 437 (11.8) | 735 (9.79)
  Cycle 8 (n=3,3,3,4) | 485 (48.1) | 573 (73.2) | 741 (32.8) | 1730 (32.6)

ADVERSE EVENTS:
Time Frame: Through final cut off in November 2013
Description: For frequency counts by preferred term, multiple occurrences of the same adverse event (AE) in an individual are counted only once.
Groups:
- Safety Population: Safety-Evaluable Participants
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 46/134
Other Adverse Events (participants affected / at risk) | 123/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=134)
Anaemia (Blood and lymphatic system disorders) | 2
Aplasia pure red cell (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiorespiratory arrest (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 4
Bacteraemia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Colonic abscess (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Pneumococcal infection (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 8
Tooth avulsion (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Tumour lysis sydrome (Metabolism and nutrition disorders) | 4
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=134)
Lymphopenia (Blood and lymphatic system disorders) | 19
Anaemia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 35
Pyrexia (General disorders) | 13
Oedema peripheral (General disorders) | 12
Fatigue (General disorders) | 7
Bronchitis (Infections and infestations) | 15
Nasopharyngitis (Infections and infestations) | 15
Infusion related reaction (Injury, poisoning and procedural complications) | 107
Weight decreased (Investigations) | 10
Decreased appetite (Metabolism and nutrition disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 8
Insomnia (Nervous system disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9

LIMITATIONS AND CAVEATS:
Pharmacodynamic results were limited because number of participants was inversely proportional to length of follow-up. In other words, there were fewer participants still in the trial as the follow-up period became longer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.